CLINICAL TRIAL: NCT03088761
Title: Changes in the Cuff Pressure in Infants in the Absence of Nitrous Oxide
Brief Title: Cuff Pressure in Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul Science University (Other)
Responsible Party: Principal Investigator, Kemal Tolga Saracoglu, Associate Professor MD, Istanbul Science University
Other Study IDs: 44140529
Record Dates: First submitted 2017-03-18; First posted 2017-03-23 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Myelomeningocele; Prone Position
Keywords: tracheal tube; cuff pressure
MeSH Terms: conditions — Meningomyelocele

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- cuffed tube pressure group: The pressures of cuffed tracheal tubes will be monitored simultaneously with a cuff manometer and pressure transducer. The measurements will be observed continuously. When the cuff pressure is noted to exceed 15 cmH2O, the cuff will be deflated immediately to less than 15 cmH2O. The time when the correction occurred, the time interval between corrections and the number of corrections during surgery will be recorded.
  The baseline cuff pressure will be assessed in the supine position after which time a second measurement will be made in the prone position. A blind investigator will check and record the findings of cuffed tracheal tube.
  Interventions: Device: cuffed tracheal tube

INTERVENTIONS:
Device: cuffed tracheal tube — the changes in cuff pressure will be determined using a cuff manometer

SUMMARY:
The changes in the cuff pressure in the absence of nitrous oxide are less clear.In the current study, we aim to determine the changes in cuff pressure over time in infants undergoing myelomeningocele repair in prone position under general anesthesia in the absence of N2O.

DETAILED DESCRIPTION:
Introduction:

During perioperative period some factors may change the endotracheal tube (ETT) cuff pressure. They include time (1), changes in core temperature (2), neuromuscular blockade (3), sedation (4), altitude (5), use of nitrous oxide (6,7), changes in tracheal muscle tone and respiratory system impedance (8), different body, head and neck positions (9), mechanical ventilation and transoesophageal echocardiography probe insertion (10).

Some have chosen to avoid the use of nitrous oxide (N2O) during surgery because of the theoretical risk of multiple deleterious effects on the neurologic, cardiovascular, hematologic and immune systems. In addition, N2O diffuses into all gas-filled cavities increasing their sizes and pressures including ETT cuffs (11). ETT cuff pressure increases after exposure to nitrous oxide (12).

However, the changes in the cuff pressure in the absence of nitrous oxide are less clear. Kako et al. (13) investigated the relationship between head and neck position and ETT cuff pressure in children in the absence of N2O in the supine position. In this study, 1000 intracuff readings were evaluated in 200 children based on position of the head and neck. They found that cuff pressure increased in two-thirds of the measurements 545 out of 1000 when compared with the neutral position. Most frequently change was noted with neck flexion. The mean increase in cuff pressure was 7.2±8.3 cmH2O from the neutral position (p<0.05).

In the current study, we aim to determine the changes in cuff pressure over time in infants undergoing myelomeningocele repair in prone position under general anesthesia in the absence of N2O.

Methods:

This prospective observational study was approved by the Institutional Review Board of Istanbul Science University. After parents are given a detailed explanation about of the procedure of ETT placement for general anesthesia, consent for their children's participation will be sought. The study will be registered at ClinicalTrials.gov.

Twenty infants undergoing repair of myelomeningocele will be recruited. Their airways will be secured with a cuffed ETT. All infants will undergo surgery in the prone position.

Anesthesia will be induced with a combination of oxygen, air, sevoflurane, intravenous remifentanil and rocuronium. After tracheal intubation with a high volume low pressure cuffed ETT (Nextech®, Istanbul, Turkey), the cuff will be inflated until there is no audible gas leak. The observer will check the gas leak using a stethoscope guided inflation over the trachea while holding continuous positive airway pressure of 20-25 cm H2O (14).

The ETT cuff pressures will be monitored simultaneously with a cuff manometer and pressure transducer (15). The measurements will be observed continuously. When the cuff pressure is noted to exceed 15 cmH2O, the cuff will be deflated immediately to less than 15 cmH2O. The time when the correction occurred, the time interval between corrections and the number of corrections during surgery will be recorded.

The baseline cuff pressure will be assessed in the supine position after which time a second measurement will be made in the prone position. A blind investigator will check and record the cuff pressure. If the pressure is between 10-15 cmH2O, no intervention will be performed. If the pressure exceeds 15 cmH2O, the cuff pressure will be managed as described above. The cuff pressures will be compared over time within patients. In addition, heart rate, end-tidal CO2, temperature and peak airway pressure will be recorded every 15 min.

Statistics:

All data that are normally distributed will be summarized as means ± standard deviation. Data that are not normally distributed will be summarized as medians and 25-75th percentile. Cuff pressure and all other interval data that will be measured over time will be analyzed using repeated-measures ANOVA with the Tukey (or Dunnett) post-hoc test. Comparing supine and prone positions, cuff pressures will be analyzed using two-way repeated measures ANOVA. Baseline demographic data will be compared using unpaired t-test for normally distributed data and Mann Whitney U test for data that are not normally distributed. P<0.05 will be accepted.

ELIGIBILITY:
Inclusion Criteria:

* male and female infants undergoing meningomyelocele repair

Exclusion Criteria:

* tracheal intubation with uncuffed tube, the use of N2O during anesthesia, accompanying disease like hydrocephalus

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 1-30 days old infants undergoing meningomyelocele repair
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2017-09-30 (Estimated); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
the change in cuff pressure | four months
  the change in cuff pressure will be recorded during prone position

CONTACTS AND LOCATIONS:
Overall Officials: Kemal T Saracoglu, Principal Investigator — Istanbul Science University School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Motoyama A, Asai S, Konami H, Matsumoto Y, Misumi T, Imanaka H, Nishimura M. Changes in endotracheal tube cuff pressure in mechanically ventilated adult patients. J Intensive Care. 2014 Jan 31;2(1):7. doi: 10.1186/2052-0492-2-7. eCollection 2014. PMID 25520824
- [Result] Kako H, Alkhatib O, Krishna SG, Khan S, Naguib A, Tobias JD. Changes in intracuff pressure of a cuffed endotracheal tube during surgery for congenital heart disease using cardiopulmonary bypass. Paediatr Anaesth. 2015 Jul;25(7):705-10. doi: 10.1111/pan.12631. Epub 2015 Mar 4. PMID 25735902
- [Result] Lizy C, Swinnen W, Labeau S, Poelaert J, Vogelaers D, Vandewoude K, Dulhunty J, Blot S. Cuff pressure of endotracheal tubes after changes in body position in critically ill patients treated with mechanical ventilation. Am J Crit Care. 2014 Jan;23(1):e1-8. doi: 10.4037/ajcc2014489. PMID 24382623
- [Result] Nseir S, Brisson H, Marquette CH, Chaud P, Di Pompeo C, Diarra M, Durocher A. Variations in endotracheal cuff pressure in intubated critically ill patients: prevalence and risk factors. Eur J Anaesthesiol. 2009 Mar;26(3):229-34. doi: 10.1097/eja.0b013e3283222b6e. PMID 19244697
- [Result] Orsborn J, Graham J, Moss M, Melguizo M, Nick T, Stroud M. Pediatric Endotracheal Tube Cuff Pressures During Aeromedical Transport. Pediatr Emerg Care. 2016 Jan;32(1):20-2. doi: 10.1097/PEC.0000000000000365. PMID 25834962
- [Result] Beydon L, Gourgues M, Talec P. [Endotracheal tube cuff and nitrous oxide: bench evaluation and assessment of clinical practice]. Ann Fr Anesth Reanim. 2011 Sep;30(9):679-84. doi: 10.1016/j.annfar.2011.03.017. Epub 2011 Jun 25. French. PMID 21705180
- [Result] Tu HN, Saidi N, Leiutaud T, Bensaid S, Menival V, Duvaldestin P. Nitrous oxide increases endotracheal cuff pressure and the incidence of tracheal lesions in anesthetized patients. Anesth Analg. 1999 Jul;89(1):187-90. doi: 10.1097/00000539-199907000-00033. PMID 10389801
- [Result] Plotnikow GA, Roux N, Feld V, Gogniat E, Villalba D, Ribero NV, Sartore M, Bosso M, Quiroga C, Leiva V, Scrigna M, Puchulu F, Distefano E, Scapellato JL, Intile D, Planells F, Noval D, Bunirigo P, Jofre R, Nielsen ED. Evaluation of tracheal cuff pressure variation in spontaneously breathing patients. Int J Crit Illn Inj Sci. 2013 Oct;3(4):262-8. doi: 10.4103/2229-5151.124148. PMID 24459624
- [Result] Godoy AC, Vieira RJ, Capitani EM. Endotracheal tube cuff pressure alteration after changes in position in patients under mechanical ventilation. J Bras Pneumol. 2008 May;34(5):294-7. doi: 10.1590/s1806-37132008000500008. English, Portuguese. PMID 18545825
- [Result] Tan PH, Lin VC, Chen HS, Hung KC. The effect of transoesophageal echocardiography probe insertion on tracheal cuff pressure. Anaesthesia. 2011 Sep;66(9):791-5. doi: 10.1111/j.1365-2044.2011.06789.x. Epub 2011 Jun 24. PMID 21707563
- [Result] Tobias JD. Applications of nitrous oxide for procedural sedation in the pediatric population. Pediatr Emerg Care. 2013 Feb;29(2):245-65. doi: 10.1097/PEC.0b013e318280d824. PMID 23546436
- [Result] Maino P, Dullenkopf A, Bernet V, Weiss M. Nitrous oxide diffusion into the cuffs of disposable laryngeal mask airways. Anaesthesia. 2005 Mar;60(3):278-82. doi: 10.1111/j.1365-2044.2004.04072.x. PMID 15710013
- [Result] Kako H, Krishna SG, Ramesh AS, Merz MN, Elmaraghy C, Grischkan J, Jatana KR, Ruda J, Tobias JD. The relationship between head and neck position and endotracheal tube intracuff pressure in the pediatric population. Paediatr Anaesth. 2014 Mar;24(3):316-21. doi: 10.1111/pan.12308. Epub 2013 Nov 18. PMID 24238105
- [Result] Grant T. Do current methods for endotracheal tube cuff inflation create pressures above the recommended range? A review of the evidence. J Perioper Pract. 2013 Dec;23(12):292-5. doi: 10.1177/175045891302301205. PMID 24404708
- [Result] Krishna SG, Ramesh AS, Jatana KR, Elmaraghy C, Merz M, Ruda J, Tobias JD. A technique to measure the intracuff pressure continuously: an in vivo demonstration of its accuracy. Paediatr Anaesth. 2014 Sep;24(9):999-1004. doi: 10.1111/pan.12437. Epub 2014 May 24. PMID 24860935